CLINICAL TRIAL: NCT00253838
Title: A Randomized Controlled Trial Comparing a Titanium to a Cobalt Chrome Femoral Stem in Revision Hip Arthroplasty: A Pilot Study
Brief Title: A Comparison of Two Type of Stems in Revision Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OHREB 2001215-01H
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Hip Arthroplasty
Keywords: revision hip arthroplasty; bone mineral density

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restoration HA Stem (Active Comparator): The Restoration hip stem, is made from titanium alloy, a different type of metal that has a roughened surfacing and allows for a hydroxylapatite (HA) coating
  Interventions: Procedure: Restoration HA stem
- Solution stem (Sham Comparator): The Solution stem is made from Cobalt Chrome, a type of metal, and does not have a hydroxylapatite (HA) coating.
  Interventions: Procedure: Solution stem

INTERVENTIONS:
Procedure: Restoration HA stem — The Restoration hip stem, is made from titanium alloy, a different type of metal that has a roughened surfacing and allows for a hydroxylapatite (HA) coating to be applied to the entire length of the stem.
  Other Names: non applicable
  Arms: Restoration HA Stem
Procedure: Solution stem — The Solution stem is made from Cobalt Chrome, a type of metal, and does not have a hydroxylapatite (HA) coating.
  Other Names: non applicable
  Arms: Solution stem

SUMMARY:
This study compares two different hip stem components. Both hip stems used in this study allow the femur bone to attach and grow into them for stability. The main difference between the two stems is that one of the stems, the Solution® Stem, is made from Cobalt Chrome, a type of metal, and does not have a hydroxylapatite (HA) coating, while the second stem included in the study, the Restoration hip stem, is made from titanium alloy, a different type of metal that has a roughened surface and allows for a hydroxylapatite (HA) coating to be applied to the entire length of the stem. The HA coating is a thin calcium phosphate layer on the stem to encourage the bone to grow into it. We are trying to see if there is any difference in the initial bony ingrowth between the two stems and to compare the results in patients over the first two years after the surgery and then again at the five-year period.

DETAILED DESCRIPTION:
Revision total hip arthroplasty is becoming increasingly common due to the large number of primary total hip arthroplasties being performed annually. Failure of these arthroplasties has led to an increasing number of patients requiring revision arthroplasty. Various methods have been used to reconstruct the hip during a revision procedure. These have generally consisted of a cemented or uncemented femoral stem. It is now generally accepted that uncemented femoral stems have improved results over cemented stems, especially in those cases with compromised bone stock. There are two main alloys used for the femoral revision component, that is cobalt chrome and titanium. There may be certain advantages to the use of titanium, in particular, a reduction in future bone loss caused by stress shielding. Stress shielding is commonly seen with cobalt chrome implants. In order to assess this and the overall survival of these two different implants a randomized clinical trial is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for revision hip arthropathy

Exclusion Criteria:

* Under 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2001-10; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety of surgical implant | 24 months
  Safety of surgical implant will be assessed by reviewing revision rates and complication rates post surgery

SECONDARY OUTCOMES:
Patient outcome measures | pre-op, 6, 12, 24, 60 months
  Patient outcome measures will be assessed using the SF-12 and WOMAC questionnaires.
Effectiveness of surgical implant | 24 months
  The Harris Hip Score will be used to evaluate the effectiveness of the surgical implant

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Kim, MD, FRCSC, Principal Investigator — OHRI
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada